CLINICAL TRIAL: NCT04928378
Title: Management of Osteoarticular Infection Due to Multidrug Resistant Mycobacterium Tuberculosis Strains in France
Brief Title: Bone Resistant Tuberculosis
Acronym: TboneR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210051
Record Dates: First submitted 2021-05-21; First posted 2021-06-16 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-01

CONDITIONS: Bone and Osteoarticular Infection Due to MDR M. Tuberculosis Strains
Keywords: Mycobacterium tuberculosis; Multi drug resistance; Bone; osteoarticular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Descriptive retrospective study — characterization of the diagnosis, management and outcome of patients with osteoarticular infection due to MDR M. tuberculosis in France (MDR IOATB).

SUMMARY:
The recommendations for the treatment of MDR tuberculosis are based on pulmonary tuberculosis since there is a lack of specific recommendations for TB bone and osteoarticular disease, including those due to multi drug resistance strains (MDR IOATB). Given the lack of data regarding MDR IOATB, it may be helpful to study the diagnosis, medical treatment, surgical indications and prognosis of a cohort of MDR IOATB patients.

DETAILED DESCRIPTION:
Due to the lack, in the guidelines regarding bone and osteoarticular infections due to MDR M. tuberculosis strains, this study aims to characterize the diagnosis, management and outcome of patients with osteoarticular infection due to MDR M. tuberculosis in France (MDR IOATB).

Aim: descriptive study of diagnosis, therapeutics and outcome of patients with bone and osteoarticular infection with MDR IOATB in France.

Set up: patients registered in the database of the National Reference Center (CNR) for MDR IOATB in France, treated for MDR IOATB between January 1, 2007 and December 31, 2018 will be included and analyzed.

Study design: retrospective study on historical cohort

ELIGIBILITY:
Inclusion Criteria:

* Any patient with an MDR IOATB whose sample and / or strain has been referred to the National Reference Center (CNR) for mycobacteria in France, will be included.

Exclusion Criteria:

* Patient refusing to have their data used.
* Patients under guardianship or curators, patients under legal protection will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered in the database of the National Reference Center (CNR) for MDR IOATB in France, treated for MDR IOATB between January 1, 2007 and December 31, 2018 will be included and analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
study of infected population with MDR TB IOATB | Through study completion, an average of 1 year
  Description of patients with MDR IOATB on anamnestic, clinical, paraclinical, diagnosis, prognosis, therapeutic and outcome level.
  Data collected for : demographics (age, sex), history of previous treatment for tuberculosis (list of), immunocompromised status (and which kind), clinical presentation, tuberculosis localization, administered treatment (sort, duration), adverse events (number of patients with treatment-related adverse events using WHO scale), surgery (y or n and which surgery: descriptive) and treatment outcomes death, cure, relapse, lost in follow up)

SECONDARY OUTCOMES:
Drug susceptibility testing | Through study completion, an average of 1 year
  Testing for phenotypic drug susceptibility using the proportion method and genetic mutations involved in antituberculosis drug resistance identified with biomolecular tool.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Aubry, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided